CLINICAL TRIAL: NCT01368380
Title: Hand in Hand. Psychological Intervention for Breast Cancer Patients and Their Partners. A Randomised, Controlled Trial.
Brief Title: Hand in Hand. Psychological Support and Counseling to Breast Cancer Patients and Their Partners
Acronym: HIH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Collaborators: Odense University Hospital (Other); Ringsted Hospital (Unknown); University of Copenhagen (Other); Region of Southern Denmark (Other); Danish Cancer Society (Other)
Responsible Party: Principal Investigator, Anne Nicolaisen, MPH, Ph.D. student, University of Southern Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NFK-SDU-2011-5
Record Dates: First submitted 2011-05-23; First posted 2011-06-07 (Estimated); Last update posted 2015-02-26 (Estimated); Status verified 2015-02

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Partners; Couples; Attachment; Intervention
MeSH Terms: conditions — Breast Neoplasms | interventions — Psychosocial Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Psychological Intervention (Experimental)
  Interventions: Behavioral: Psychological intervention
- Usual care (No Intervention)

INTERVENTIONS:
Behavioral: Psychological intervention — Couples in the intervention group attends six to eight couple-sessions performed by a psychologist.
  Arms: Psychological Intervention

SUMMARY:
This study evaluates the effect of a psychological intervention to breast cancer patients and their partners compared to a control group receiving usual care

DETAILED DESCRIPTION:
The intervention intends to improving the patient and partners well-being, quality of life and their relationship adjustment.

The couples in the intervention group participates i six to eight couple sessions. The sessions is conducted by an experienced psychologist and takes place one to five months after the patients cancer diagnosis. The control group receives usual care.

The framework of the intervention is attachment theory and the psychologists support and advise the couples in talking candidly about their feelings regarding their new life situation with cancer. The psychologist focus on the couples ability to feel comfortable and safe in each others presence.

ELIGIBILITY:
Inclusion Criteria:

* Women newly diagnosed with a primary breast cancer (in the last 4 weeks)
* Women cohabiting with a male partner in a romantic relationship
* Patient and partner speaks and reads danish

Exclusion Criteria:

* Patients having a previous cancer diagnosis
* Neoadjuvant therapy for breast cancer
* Previous hospital admission with diagnosed psychotic episodes

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2011-10; Primary Completion 2013-08 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Change in Impact of Event Scale (IES) | Baseline, 2 weeks post-intervention, 10 months follow-up
  IES assesses traumatic reactions to the breast cancer diagnosis. Assessed by both patients and partners
Change in The Hospital Anxiety and Depression Scale (HADS) | Baseline, 2 weeks post-intervention, 10 months follow-up
  Assesses feelings of anxiety and depressive symptoms. Assessed by both patients and partners.
Change in The Profile of Mood States - Short Form (POMS-SF) | Baseline, 2 weeks post-intervention, 10 months follow-up
  Assesses mood changes. Assessed by both patients and partners

SECONDARY OUTCOMES:
Change in Dyadic Adjustment Scale - Revised (DAS-R) | Baseline, 2 weeks post-intervention, 10 months follow-up
  Assesses relationship functioning and marital satisfaction. Assesed by both patients and partners
Change in Relationship Questionnaire (RQ) | Baseline, 2 weeks post-intervention, 10 months follow-up
  RQ provides a profile of an individual's attachment feelings and behaviour. Assessed by both patients and partners
Change in Functional Assessment of Cancer Therapy - Breast (FACT-B) | Baseline, 2 weeks post-intervention and 10 months follow-up
  Assesses health-related quality of life with additional questions for women dignosed with breast cancer.
Change in Functional Assessment of Cancer Therapy - general population (FACT-GP) | Baseline, 2 weeks post-intervention and 10 months follow-up
  Assesses health-related quality of life. Assessed by partners
Change in Functional Assessment of Chronic Illness Therapy-Fatigue | Baseline, 2 weeks post-intervention and 10 months follow-up
  Assesses individual fellings of fatigue. Assessed by the patients
Change in Post Traumatic Growth Inventory | 2-weeks post-intervention and 10 months follow-up
  Assesses positive changes in individuals experiencing traumatic life events. Assessed by both patients and partners
Change in EuroQol-5 Dimensions (EQ-5D) | Baseline, 2 weeks post-intervention and 10 months follow-up
  Assesses health-related quality of life. Assessed by both patients and partners

CONTACTS AND LOCATIONS:
Overall Officials: Dorte G Hansen, PhD, Principal Investigator — University of Southern Denmark; Mariët Hagedoorn, Professor, Study Chair — University of Groningen; Christoffer Johansen, Professor, Study Chair — Danish Cancer Society; Henrik Flyger, MD, Ph. D, Study Chair — University of Copenhagen
Locations (3):
- Denmark (3):
  - Herlev University Hospital, Herlev
  - Odense University Hospital, Odense
  - Ringsted Hospital, Ringsted

REFERENCES:
- [Derived] Nicolaisen A, Hansen DG, Hagedoorn M, Flyger HE, Rottmann N, Nielsen P, Soe K, Pedersen AE, Johansen C. Attachment-oriented psychological intervention for couples facing breast cancer: protocol of a randomised controlled trial. BMC Psychol. 2014 Jul 14;2(1):19. doi: 10.1186/2050-7283-2-19. eCollection 2014. PMID 25815190